CLINICAL TRIAL: NCT00428415
Title: The Effect of Tesofensine on Energy Balance in Humans. A Randomised, Double-Blind, Placebo-Controlled, Parallel- Group, Single Centre Study.
Brief Title: Effect of Tesofensine on Energy Balance in Humans.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NeuroSearch A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TIPO-2
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2008-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Tesofensine

INTERVENTIONS:
Drug: Tesofensine

SUMMARY:
Purpose:

To evaluate the effect of tesofensine on energy balance

ELIGIBILITY:
Inclusion Criteria:

* Overweight to obese subjects with BMI 28 - 35 kg/m² otherwise healthy
* Males 18 to 50 years of age, extremes included
* Subjects should be able to comply with study procedures
* Subjects giving written informed consent

Exclusion Criteria:

* Use of any concomitant medication including high dose vitamins and regular OTC preparations
* Subjects who have been smokers within the last year
* Subjects with specific diseases interfering with their metabolism e.g. myxoedema, Cushing's syndrome, Type 1 diabetes mellitus, significant neurological or psychiatric illness such as epilepsy, schizophrenia, depression, eating disorders such as bulimia.
* Subjects with Type 2 diabetes mellitus are ineligible unless anti-diabetic medication was not deemed necessary by the investigator and fasting (venous or arterialized capillary full blood from finger or ear) blood glucose > 6.1 mmol/l at screening. Re-test is allowed if first measure is above inclusion value. The corresponding exclusion criteria for plasma glucose is 7.0 mmol/l
* Known hypercholesterolaemia (> 7 mmol/l).
* Known hypertriglyceridaemia (> 3 mmol/l).
* Malabsorptive intestinal disorders that can be assumed to affect the absorption of tesofensine
* Mental or psychiatric disorder based on medical history only
* Subjects with systemic infections or inflammatory diseases
* Subjects currently (within the past 2 months) known to abuse or to be dependent on any drug, including alcohol (weekly consumption > 21 units of alcohol )
* Hepatic or renal dysfunction (ASAT and/or ALAT > 2 x ULN and creatinine clearance < 30 mL/min estimated by central laboratory using Cockcroft and Gault formula, respectively)
* Special diets (e.g., vegetarian, Atkins)
* Subject should not be athletics or planning major changes in physical activity during the study to an extent that may interfere with the study outcome, as judged by the investigator
* Weight change of > 3 kg within 2 months prior to screening
* Surgically treated obesity
* History or presence of significant cardiovascular disease such as heart failure, ischemic heart disease, stroke, transient ischemic attacks
* Significant abnormalities on the ECG according to the investigators opinion. Additional exclusionary ECG values: QTcB > 450 milliseconds(ms), PR interval > 240 ms, QRS interval > 120 ms
* Hypotension (i.e. supine systolic BP < 90 mm Hg) and/or symptomatic orthostatic hypotension (clinical symptoms of orthostatic hypotension associated with a decline ≥ 20 mm Hg in systolic BP at one minute after standing compared with the previous supine systolic BP obtained after 5 minutes of quiet rest) at screening visit
* Hypertension (i.e. sitting diastolic BP ≥ 95 mm Hg and sitting systolic BP ≥ 155 mm Hg) as well as HR>90 bpm
* Known HIV infection (no tests required)
* Clinically significant or potentially disabling eye disorder, including uncontrolled glaucoma
* Serologic evidence of active hepatitis B and/or C
* History of cancer within the past 5 years, excluding treated basal cell carcinoma
* Subjects previously treated with tesofensine
* Subjects treated with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study drug

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Effect on 24-h EE (energy expenditure) after 14 days dosing, adjusted for FFM(Fat-Free Mass) and FM (Fat Mass) changes

SECONDARY OUTCOMES:
24-h fat oxidation, spontaneous physical activity, fecal excretion of energy and fat (respiratory chamber),Changes in body weight and composition
Physical Measure(Waist circumference, waist-hip ratio, change in BMI, Sagittal diameter and DEXA, Spontaneous energy intake at lunch test
Metabolic measures (Total triglycerides, Cholesterol-total, LDL-C, HDL-C, LDH, Blood glucose fasting, HbA1c, C-reactive protein, Insulin, Adiponectin, FFA, CCK, Ghrelin, and Leptin)
Data from questionnaires( Satiety & Appetite, POMS Brief)
Safety & Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Arne V Astrup, MD, Principal Investigator — Department of Human Nutrition, The Royal Veterinary & Agricultural University
Locations (1):
- NeuroSearch A/S, Ballerup Municipality, Denmark